CLINICAL TRIAL: NCT03284203
Title: Feasibility of Inpatient and At-Home Use of Handheld Spirometry (SpiroPD)
Brief Title: Feasibility of At-Home Handheld Spirometry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The aims represented in this study are also included in another, larger study of at-home COPD care. There was insufficient research team support to complete both protocols and the work would have been duplicative. Thus, we have terminated this study.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB17-0562
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SpiroPD (Experimental): Participants in the intervention arm will be given a handheld spirometry device to take home and use daily for 30 consecutive days.
  Interventions: Device: SpiroPD

INTERVENTIONS:
Device: SpiroPD — At the time of their initial study visit, study participants will be given a SpiroPD device for use at home following instruction in the hospital or clinic. Patient adherence to daily testing over one-month will be monitored using real-time capture Wi-Fi-data from the SpiroPD data portal.

SUMMARY:
The investigators' central hypotheses predict that the handheld spirometry device will be feasible for inpatient and at-home use, and is equally efficacious at determining lung function when compared to traditional, bedside spirometry measurements. To test these hypotheses, the investigators propose the following specific aims:

Specific Aim 1: Determine the correlation of SpiroPD handheld spirometry measurements with bedside Koko spirometry lung function.

Hypothesis: Correlation between the two lung function tests will be substantial for both hospitalized and ambulatory patients.

Specific Aim 2: To determine the feasibility, adherence, and preliminary management efficacy of home SpiroPD testing.

Hypotheses: (1) Patients will demonstrate substantial adherence to daily home spirometry testing; (2) medication adherence will increase significantly in patients who are adherent to daily home spirometry testing; (3) acute care utilization will decrease significant in adherent patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) results in nearly 750,000 hospitalizations annually and is the third leading cause of "early" (within 30-day) hospital readmissions in the United States. Curbing preventable early readmissions for acute exacerbations of COPD (AECOPD) has become a national priority, as demonstrated by the Medicare Hospital Readmissions Reduction financial penalty program. One critical barrier in assessing readmission risk is the lack of an easily-measured 'vital sign' for COPD: accurate, timely measurements of lung function. Unlike other medical problems that have validated, easily-obtained measurements of organ function, COPD evaluation often defaults to patient report and physician evaluation without critical physiologic data. This lack of objective pulmonary function data during AECOPD in turn leads to critical errors in disease severity assessment. However, the required, repeated measurements by spirometry that can demonstrate responses to therapy can be time-consuming and expensive to perform in a laboratory, and both equipment and staffing infrastructure for bedside testing is cumbersome and often not prioritized. For these reasons, spirometry frequently is not done for patients with AECOPD.

To monitor patient responses to therapy and to assess risks based on objective measures, the investigators propose to the study the use of a portable, patient-driven device ("SpiroPD") that can be used in both in-patient and outpatient settings, and that reports (via the internet) values collected in real time. While the device has been used in the lung transplant community and for patients with cystic fibrosis, no studies have been done to validate its use in COPD. This protocol involves in-hospital patient training with the device followed by serial measurements at home in the first 30 days post hospital-discharge.

Demonstration in a pilot, single-center trial of the usefulness of real-time, repeated hand-held spirometry to provide objective measurements of lung function in AECOPD will have a substantial impact on both patient health outcomes and on health care utilization and will set the stage for appropriate next-step studies and NIH grant applications. It is unknown whether this specific technology will be acceptable in the target population, though previous research suggests that older patients may be more willing to use home monitoring technology. This multi-disciplinary research team includes providers from the Department of Medicine and the UCM COPD Readmissions Program team.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years
* Physician-diagnosed COPD
* Able to perform spirometry
* Access to wireless internet at home
* Visual acuity of at least 20/50 in one eye

Exclusion Criteria:

* Currently in ICU
* Physician declines to provide consent
* Patient unable to provide consent or declines to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Press, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from September to December 2017 at the University of Chicago Medical Center.
Pre-assignment Details: No participants were excluded from the study except those who did not meet the eligibility criteria.
Period: Overall Study
Arm/Group | SpiroPD
Started | 8
Completed | 5
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | SpiroPD
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.85 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Measure of race and ethnicity of participants
  Participants
    Race/Ethnicity: White | 1
    Race/Ethnicity: Black/African American | 7
    Race/Ethnicity: Asian | 0
    Race/Ethnicity: American Indian/Alaskan Native | 0
    Race/Ethnicity: Native Hawaiian/Other Pacific Islander | 0
    Race/Ethnicity: Hispanic/Latino | 0
    Race/Ethnicity: Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Comparison of KOKO Spirometry to SpiroPD Use
Description: Participants will use the handheld spirometry device every day for 30 days. After use, the device will store spirometry measurements for each patient each day and the data will be synced over wifi to each individual's associated online account. Daily measurements from the SpiroPD device will be collected over the course of 30 days. These measurements will then be compared against spirometry measurements collected using the bedside KoKo machine during baseline and 30-day follow-up visits.
Time Frame: 30 days from patient enrollment
Population: We have reported data from baseline KOKO spirometry measurements vs. in-hospital SpiroPD use. However, none of the 8 enrolled participants used the SpiroPD device at home and thus, no data from at-home spirometry exists for this analysis.
Measure: Mean (Standard Deviation); unit: percentage of FVC
Arm/Group | SpiroPD
Number analyzed (Participants) | 8
percentage of FVC
  FVC % Predicted KOKO | 57.01 (22.83)
  FVC % Predicted Baseline SpiroPD | 64.33 (24.15)
  FVC % Predicted at-home SpiroPD: number analyzed (Participants) | 0

2. Secondary Outcome: Adherence to Using the SpiroPD Device at Home on a Daily Basis
Description: Daily use of the SpiroPD will be measured by way of captured spirometry measurements. If there is no recorded spirometry measurement in the SpiroPD device for certain days, those days will be considered when discussing non-adherence to daily use of the SpiroPD.
Time Frame: 30 days from patient enrollment
Population: None of the 8 enrolled participants adhered to using the SpiroPD at home. No at-home data was able to be collected during this study; thus, there are no results to report.
Arm/Group | SpiroPD
Number analyzed (Participants) | 0

3. Secondary Outcome: Feasibility of Patients to Use the SpiroPD Device at Home Consistently
Description: Feasibility, or ease of use, will be measured by tracking the number of inquiries received on the designated SpiroPD help line. Each inquiry will be measured and tracked using an inquiry intake form. The type of inquiry or issue the patient is having and the possible solutions to the issue will be recorded. The patient's study ID and the date and time of their call will be recorded. These metrics along with adherence measurements will be factored in when discussing the feasibility of the SpiroPD device.
Time Frame: 30 days from patient enrollment
Population: There were no inquiries received on the SpiroPD help line. Thus, there is no data to report regarding the feasibility of SpiroPD.
Arm/Group | SpiroPD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed over 30 days post hospital discharge after enrollment into this study.
Description: Any serious negative health outcome, such as mortality.
Arm/Group | SpiroPD
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03284203/Prot_SAP_002.pdf
  • Informed Consent Form (2018-04-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03284203/ICF_003.pdf